CLINICAL TRIAL: NCT04596631
Title: Efficacy and Safety of Oral Semaglutide Versus Placebo Both in Combination With Metformin and/or Basal Insulin in Children and Adolescents With Type 2 Diabetes
Brief Title: A Research Study to Compare a New Medicine Oral Semaglutide to a Dummy Medicine in Children and Teenagers With Type 2 Diabetes
Acronym: PIONEER TEENS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9924-4437; U1111-1218-1527 (Other: World Health Organization (WHO)); 2018-002952-34 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide - max. tolerated dose (Experimental): Participants will receive semaglutide tablets once daily in addition to background treatment with metformin or basal insulin or both, in addition to diet and exercise.
  Interventions: Drug: Oral semaglutide
- Placebo (semaglutide) (Placebo Comparator): Participants will receive semaglutide placebo tablets once daily in addition to background treatment with metformin or basal insulin or both, in addition to diet and exercise.
  Interventions: Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Oral semaglutide — Oral semaglutide treatment for 52 weeks. All participants will be dose-escalated to an individual maximum tolerated dose.
  Arms: Semaglutide - max. tolerated dose
Drug: Placebo (semaglutide) — Placebo treatment for 52 weeks.
  Arms: Placebo (semaglutide)

SUMMARY:
This study compares 2 medicines for type 2 diabetes: semaglutide (new medicine) and a dummy medicine (placebo). Semaglutide will be tested to see how well it works compared to the dummy medicine. The study will also test if semaglutide is safe in children and teenagers. Participants will either get semaglutide or the dummy medicine - which one is decided by chance. Participants will take 1 tablet of the study medicine every morning on an empty stomach. They have to wait 30 minutes before they eat, drink or take any other medication by mouth. The study will last for about 1 year and 3 months (66 weeks). Participants will have 12 clinic visits and 8 phone calls with the study doctor. At all 12 clinic visits, participants will have blood samples taken. Participants will also be asked some questions.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from parent(s) or legally acceptable representative (LAR) and child assent from the subject obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
* Male or female, aged 10 to below 18 years at the day of randomisation
* HbA1c 6.5%-11.0% (47-97 mmol/mol) (both inclusive)
* Diagnosed with type 2 diabetes mellitus according to the American Diabetes Association criteria and treated with:
* stable metformin dose (stable metformin dose is defined as at least 1000 mg daily or the maximum tolerated dose for 56 days or longer prior to screening) or
* stable metformin dose and a stable dose of basal insulin (stable dose of basal insulin is defined as basal insulin treatment equal to or more than 30 days prior to screening, compared to the dose at screening, dose adjustments of ± 25% are allowed) or
* stable dose of basal insulin

Exclusion Criteria:

* Diagnosis of type 1 diabetes
* Maturity onset diabetes of the young (MODY)
* Positive insulinoma associated-protein 2 (IA-2) antibodies or anti-glutamic acid decarboxylase (anti-GAD) antibodies.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in glycosylated haemoglobin (HbA1c) | Week 0, week 26
  Percentage point

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose (FPG) | Week 0, week 26
  mmol/L
Change from baseline in body mass index (BMI) standard deviation score (SDS) | Week 0, week 26
  SDS
Change from baseline in glycosylated haemoglobin (HbA1c) | Week 0, week 52
  Percentage point
Change from baseline in FPG | Week 0, week 52
  mmol/L
Change from baseline in body weight | Week 0, week 26
  kg
Change from baseline in body weight | Week 0, week 52
  kg
Relative change from baseline in body weight | Week 0, week 26
  Percentage
Relative change from baseline in body weight | Week 0, week 52
  Percentage
Change from baseline in waist circumference | Week 0, week 26
  cm
Change from baseline in waist circumference | Week 0, week 52
  cm
Change from baseline in BMI SDS | Week 0, week 52
  SDS
BMI percentile (age and gender adjusted) | Week 0, week 26
  Percent
BMI percentile (age and gender adjusted) | Week 0, week 52
  Percent
Change from baseline in systolic blood pressure | Week 0, week 26
  mmHg
Change from baseline in systolic blood pressure | Week 0, week 52
  mmHg
Change from baseline in diastolic blood pressure | Week 0, week 26
  mmHg
Change from baseline in diastolic blood pressure | Week 0, week 52
  mmHg
HbA1c below 7.0% (53 mmol/mol) (yes/no), American Diabetes Association (ADA) target and International Society for Pediatric and Adolescent Diabetes (ISPAD) guidelines from 2018 | At week 26
  Count of participants
HbA1c equal to or below 6.5% (48 mmol/mol) (yes/no), American Association of Clinical Endocrinologists (AACE) target | At week 26
  Count of participants
HbA1c below 7.0% (53 mmol/mol) (yes/no), ADA target and ISPAD guidelines from 2018 | At week 52
  Count of participants
HbA1c equal to or below 6.5% (48 mmol/mol) (yes/no), AACE targetat week 26 | At week 52
  Count of participants
Time to additional anti-diabetic medication (to support the treatment policy estimand) | Week 0 - week 52
  Days
Time to rescue medication (to support the hypothetical estimand) | Week 0 - week 52
  Days
Number of treatment-emergent adverse events (TEAEs) during exposure to trial product | Week 0 - week 57
  Count of events
Number of treatment-emergent severe or blood glucose confirmed symptomatic hypoglycaemic episodes | From randomisation (week 0) to week 26
  Count of episodes
Number of treatment-emergent severe or blood glucose confirmed symptomatic hypoglycaemic episodes during exposure to trial product | Week 0 - week 57
  Count of episodes
Treatment emergent severe or blood glucose confirmed symptomatic hypoglycaemia episode | From randomisation (week 0) to week 26
  Count of participants
Treatment-emergent severe or blood glucose confirmed symptomatic hypoglycaemia episode during exposure to trial product | Week 0 - week 57
  Count of participants
Change from baseline in amylase | Week 0, week 26
  U/L
Change from baseline in amylase | Week 0, week 52
  U/L
Change from baseline in lipase | Week 0, week 26
  U/L
Change from baseline in lipase | Week 0, week 52
  U/L
Change from baseline in insulin-like growth factor 1 (IGF-1) | Week 0, week 26
  ng/mL
Change from baseline in insulin-like growth factor 1 (IGF-1) | Week 0, week 52
  ng/mL
Change from baseline in insulin-like growth factor binding protein 3 (IGFBP 3) | Week 0, week 26
  ng/mL
Change from baseline in insulin-like growth factor binding protein 3 (IGFBP 3) | Week 0, week 52
  ng/mL
Change from baseline in calcitonin | Week 0, week 26
  pmol/L
Change from baseline in calcitonin | Week 0, week 52
  pmol/L
Change from baseline in estradiol (for girls) | Week 0, week 26
  pmol/L
Change from baseline in estradiol (for girls) | Week 0, week 52
  pmol/L
Change from baseline in testosterone (for boys) | Week 0, week 26
  nmol/L
Change from baseline in testosterone (for boys) | Week 0, week 52
  nmol/L
Change from baseline in prolactin | Week 0, week 26
  mIU/L
Change from baseline in prolactin | Week 0, week 52
  mIU/L
Change from baseline in thyroid stimulating hormone (TSH/thyrotropin) | Week 0, week 26
  mIU/L
Change from baseline in thyroid stimulating hormone (TSH/thyrotropin) | Week 0, week 52
  mIU/L
Change from baseline in follicle stimulating hormone (FSH) | Week 0, week 26
  mIU/mL
Change from baseline in follicle stimulating hormone (FSH) | Week 0, week 52
  mIU/mL
Change from baseline in luteinizing hormone (LH) | Week 0, week 26
  mIU/mL
Change from baseline in luteinizing hormone (LH) | Week 0, week 52
  mIU/mL
Change from baseline in dehydroepiandrosterone sulfate (DHEAS) | Week 0, week 26
  μmol/L
Change from baseline in dehydroepiandrosterone sulfate (DHEAS) | Week 0, week 52
  μmol/L
Anti-semaglutide antibody status | Week 0 - week 57
  Count of participants
Anti-semaglutide antibody titer | Up to 57 weeks
  Count of participants
Anti-semaglutide antibodies with in vitro neutralising effect to semaglutide | Week 0 to week 57
  Count of participants
Anti-semaglutide antibodies cross reacting with endogenous GLP-1 | Week 0 to week 57
  Count of participants
Cross reacting antibodies with in vitro neutralising effect to endogenous GLP-1 | Week 0 to week 57
  Count of participants
Height velocity | At week 26
  cm/year
Height velocity | At week 52
  cm/year
Change from baseline in height SDS | Week 0, week 26
  SDS
Change from baseline in bone age assessment, X-ray | Week 0, week 52
  Years
Change from baseline in pubertal assessment (Tanner staging) | Week 0, week 26
  Stage 1-5 where 5 is full sexual maturity
Change from baseline in pubertal assessment (Tanner staging) | Week 0, week 52
  Stage 1-5 where 5 is full sexual maturity
Change from baseline in pulse rate | Week 0, week 26
  Beats/minute
Change from baseline in pulse rate | Week 0, week 52
  Beats/minute
Change from pre-dose to post-dose (25 and 40 min) in lactate | At week 12
  mmol/L
Change from pre-dose to post-dose (25 and 40 min) in lactate | At week 26
  mmol/L
Apparent clearance (CL/F) | Week 0 - week 52
  L/h
Average concentration (Cavg) | Week 0 - week 52
  nmol/L
SNAC plasma concentrations | Week 0 - week 52
  ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (95):
- United States (23):
  - UAB Ped Endo Children's Hosp, Birmingham, Alabama
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - Yale School Of Medicine, New Haven, Connecticut
  - Nemours Chld Clnc Jacksonville, Jacksonville, Florida
  - Nemours Children's Health, Pensacola, Florida
  - University of South Florida Diabetes Center, Tampa, Florida
  - Children's Healthcare Atlanta, Atlanta, Georgia
  - Columbus Research Foundation, Columbus, Georgia
  - Indiana Uni School of Med-Ped, Indianapolis, Indiana
  - University Of Louisville Research Foundation, Louisville, Kentucky
  - Pennington Biomed Res Ctr, Baton Rouge, Louisiana
  - Barry J. Reiner, MD LLC, Baltimore, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - UBMD Peds-Div of Endo/Diabetes, Buffalo, New York
  - UPMC Child Hosp-Pittsburgh, Pittsburgh, Pennsylvania
  - Monument Health Clinical Rsrch, Rapid City, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Tech University HSC, Amarillo, Texas
  - Univ Of Texas Hlth Science Cntr, San Antonio, Texas
  - NE Clin Res of San Antonio, San Antonio, Texas
  - Pediatric Endo UVHS, Charlottesville, Virginia
  - Virginia Commonwealth University_Richmond, Richmond, Virginia
  - Virginia Commonwealth Univ, Richmond, Virginia
- Australia (6):
  - Gosford Hospital, Gosford, New South Wales
  - Westmead Children's Hospital- The Clinical Research Centre, Westmead, New South Wales
  - Women's & Children's Hospital, North Adelaide, South Australia
  - Monash Children's Hospital, Clayton, Victoria
  - Murdoch Children's Research Institute, Parkville, Victoria
  - Perth Children's' Hospital, Nedlands, Western Australia
- Universitätsklinik für Kinder und Jugendheilkunde Haus E, Salzburg, Austria
- Belgium (3):
  - UZ Brussel, Brussels
  - Cliniques Universitaires Saint-Luc - Serv. Pédiatrie, Brussels
  - CHU - UCL Namur - Site Sainte Elisabeth_Namur_1, Namur
- Czechia (2):
  - Fakultní Nemocnice Ostrava, Ostrava-Poruba
  - Masarykova nemocnice v Usti nad Labem, o.z. - Detska klinika, Ústí nad Labem
- Greece (13):
  - University Hospital of Athens ATTIKON, Athens, Attica
  - University Hospital of Athens ATTIKON, Haidari-Athens, Attica
  - Henry Dunant Hospital Center,2nd Internal Medicine Clinic, Athens
  - U.G.H. "Attikon", Pediatric Endocrinology Outpatient Clinic, Athens
  - Athens Paediatric Center, Athens
  - Iatriko Athinon (Athens Medical Canter), Athens
  - University General Hospital of Ioannina, Endocrinology, Ioannina
  - General Hospital of Lamia, Lamia
  - Univ Gen Hospital Larisa, Larissa
  - Univ Gen Hospital Larisa, Endocrinology & Metabolic Disease, Larissa
  - Pentelis Children's Hospital - Pediatric Clinic, Penteli, Athens
  - "AHEPA" University General Hospital of Thessaloniki, Thessaloniki
  - EUROMEDICA Gen Clinic The/ki, Endocrin,Metabolism,Diabetes, Thessaloniki
- India (9):
  - Endolife Specialty Hospitals, Guntur, Andhra Pradesh
  - Excel Endocrine Centre, Kolhāpur, Maharashtra
  - P D Hinduja National Hospital and Medical Research Centre, Mumbai, Maharashtra
  - All India Institute of Medical Sciences, New Dehli, New Delhi
  - Eternal Heart Care Centre, Jaipur, Rajasthan
  - Ramdev Rao Hospital, Hyderabad, Telangana
  - Dr P V Rao - Diabetes Research Centre, Hyderabad, Telangana
  - SSKM, Kolkata, West Bengal
  - Jothydev's Diabetes & Research Center, Thriruvananthapuram
- Israel (2):
  - Soroka MC - Pediatric Endocrinology, Beersheba
  - Rambam MC - Department of Pediatrics A, Haifa
- Chronic Care Center, Hazmiyeh, Lebanon
- Malaysia (4):
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Putrajaya, Putrajaya
- Consultorio de Endocrinología y Pediatría, Puebla City, Mexico
- Hôpital d'Enfants, Rabat, Morocco
- Netherlands (2):
  - Jeroen Bosch Ziekenhuis Afdeling Cardiologie, 's-Hertogenbosch
  - De Kinderkliniek, Almere Stad
- Liggins Institute, Grafton, New Zealand
- PHI University Clinic for Children's Diseases-Skopje, Skopje, North Macedonia
- Portugal (3):
  - Hospital Da Luz S.A., Lisbon
  - Unidade Local De Saude De Santa Maria E.P.E., Lisbon
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Ponce Med School Found Inc, Ponce, Puerto Rico
- Romania (4):
  - Spitalul Judetean de Urgenta Targoviste, Târgovişte, Dâmbovița County
  - Diabet Center SRL, Brasov
  - Spitalul Clinic de Urgenta pentru Copii "M.S.Curie", Bucharest
  - Emergency County Hospital Constanta, Constanța
- Russia (7):
  - Republic Children's Hospital of Ministry of Health of Udmurt, Izhevsk
  - RMAPE, Moscow
  - NSMU paediatric clinic, Novosibirsk
  - GFHI Omsk Region "Regional Children's Clinical Hospital", Omsk
  - SPSBHI City Children out-patient clinic #44, Saint Petersburg
  - Siberian State Medical University, Tomsk
  - SAHI Sverdlovsk Reg "Regional Children's Clinical Hospital", Yekaterinburg
- Taiwan (2):
  - Taipei Mackay Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou-Dept of Pediatrics, Taoyuan District
- Ukraine (7):
  - City Clinical Hospital #9 (Dnipro) - Endocrinology department, Dnipro
  - CNPE "City Clinical Hospital #9 Dnipro City Council", Dnipro
  - Kharkiv Regional Children's Clinical Hospital - Endocrinological department, Kharkiv
  - Ukrainian scientific and practical center of endocrine surgery of MOH - department of paediatric endocrinology, Kiev
  - "Verum clinic" LLC, Kyiv
  - Komisarenko Institute of Endocrinology and Metabolism of NAMSU - Department of paediatric endocrine pathology, Kyiv
  - Vinnytsia Regional Clinical Endocrinological Centre - Therapeutic department #2, Vinnytsia
- Birmingham Children's Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com